CLINICAL TRIAL: NCT06762457
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Repeat Oral Doses of MT-501 in Healthy Volunteers
Brief Title: A First-in-Human Single and Multiple Ascending Dose Study of MT-501
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mirador Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: MT-501-101; IND 174036 (Other: US FDA)
Record Dates: First submitted 2024-12-31; First posted 2025-01-07 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteers
Keywords: MT-501; Phase 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 - Single Ascending Dose (Experimental): To assess the safety and tolerability of single doses of MT-501 following oral administration.
  Interventions: Drug: MT-501
- Part 2 - Multiple Ascending Dose (Experimental): To assess the safety and tolerability of multiple doses of MT-501 following oral administration.
  Interventions: Drug: MT-501

INTERVENTIONS:
Drug: MT-501 — MT-501 Tablets

SUMMARY:
First-in-human Study to Assess the Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) with Single and Multiple Ascending Oral Doses of MT-501 in Healthy Adults.

DETAILED DESCRIPTION:
This study is the first administration of MT-501 in healthy volunteers (HV). The purpose of the study is to evaluate the safety, tolerability, and pharmacokinetics (PK) and pharmacodynamics (PD) of single and repeat oral doses of up to 8 days of MT-501 in HV. The safety, tolerability, PK, and PD data obtained from this study will inform further development of MT-501.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female (of non-childbearing potential only) between 19 and 55 years of age inclusive, at the time of signing informed consent.
2. Females must be of non-childbearing potential and must have undergone sterilization procedures, and have official documentation, at least 6 months prior to the first dose.
3. Male subjects must use highly effective forms of contraception during sexual intercourse with female partners of childbearing potential. A non-vasectomized, male subject must agree to use a condom with a chemical barrier method.
4. Continuous non-smoker who has not used tobacco or nicotine-containing products for at least 3 months prior to the first dose of drug.
5. Good general health.
6. Able to provide written informed consent and understand and comply with the requirements of the study.

Exclusion Criteria:

1. History or presence of any clinically significant organ system disease.
2. Abnormal laboratory assessments, physical exam of ECG outside the normal range that is judged by the Investigator to be clinically significant.
3. History of alcohol or drug abuse within the past 24 months.
4. Current use or history of regular tobacco, or nicotine-containing products within 3 months prior to screening.
5. Administration or use of any investigational drug or device within 30 days preceding the first does of study drug administration.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — male and female (of non-childbearing potential only)
Enrollment: 72 (Actual)
Dates: Start 2024-12-11 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure: Number of Subjects with non-SAEs and SAES | Up to 14 days post dose
  Incidence of adverse events, clinically significant laboratory abnormalities, clinically significant electrocardiogram, vital signs, and physical examination abnormalities.

CONTACTS AND LOCATIONS:
Locations (1):
- Mirador Clinical Department, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No